CLINICAL TRIAL: NCT00163059
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial To Assess The Antidepressant Effects Of The NMDA Antagonist, CP-101,606, In Patients With Treatment Refractory Major Depressive Disorder
Brief Title: The Antidepressant Effects Of The NMDA Antagonist, CP-101,606, In Patients With MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A1611006
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2006-09-22 (Estimated); Status verified 2006-09

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — traxoprodil mesylate

INTERVENTIONS:
Drug: NMDA Antagonist, CP-101,606 (traxoprodil)

SUMMARY:
To determine if the NMDA antagonist, CP-101,606, is effective for depression

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV diagnosis of MDD

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-05; Study Completion 2005-12

PRIMARY OUTCOMES:
MADRS

SECONDARY OUTCOMES:
HAM-D

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Wichita, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1611006&StudyName=The+Antidepressant+Effects+Of+The+NMDA+Antagonist%2C+CP%2D101%2C606%2C+In+Patients+With+MDD